CLINICAL TRIAL: NCT01195428
Title: Simvastatin Effect on the Incidence of Acute Lung Injury/Adult Respiratory Distress Syndrome
Brief Title: Simvastatin Effect on the Incidence of Acute Lung Injury/Adult Respiratory Distress Syndrome (ALI/ARDS)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Minimal enrollment
Sponsor: University of Oklahoma (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 15377
Record Dates: First submitted 2010-09-02; First posted 2010-09-06 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Adult Respiratory Distress Syndrome; Acute Lung Injury
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Simvastatin (Active Comparator): Simvastatin 40 mg daily.
  Interventions: Drug: Simvastatin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Simvastatin — Simvastatin 40 mg daily
  Arms: Simvastatin
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Acute Lung Injury/Acute respiratory distress syndrome (ALI/ARDS) is a serious and frequently encountered entity in modern ICUs. Sepsis remains the most common cause of ALI/ARDS and carries the worst prognosis. The disease is characterized by an intense inflammatory process. This inflammation plays a major role in the development of gas exchange abnormalities seen in the course of the disease. Statins, primarily used as lipid-lowering agents, are now known to possess anti-inflammatory, antioxidant, antithrombogenic and vascular function-restoring actions. Therefore the investigators propose to determine if Simvastatin may be useful in decreasing the incidence of this deadly syndrome in critically ill patients.

DETAILED DESCRIPTION:
Patients will be enrolled within 24 hours of ICU admission and randomized to 1 of 2 groups: Simvastatin or placebo. Patients' management will be entirely left up to the primary team, including the need for daily laboratory and imaging. In addition, there will be no restriction on the use of any medications, as deemed necessary by the primary care physician. The primary endpoint will be the incidence of ALI/ARDS. Secondary efficacy variables will be the number of days without organ or system failure, in addition to the change in IL-6, IL-8, and TNF- α. Treatment will continue until the primary endpoint is reached, the patient discharged from the ICU or the maximum duration of 2 weeks, whichever occurs first. Patients will continued to be followed for a total of 28 days, or until discharged from the hospital, whichever occurs first.

Patients randomized, in a ratio of 1:1 to either Simvastatin 40 mg PO once daily or placebo tablet once daily in a format identical to Simvastatin.

The mortality from ALI/ARDS remains significant. In the absence of effective therapy, prophylaxis in patients at risk is an important goal to achieve. Therefore, if Simvastatin is found to decrease the incidence of ALI/ARDS, it would be a significant advance in the management of this deadly and frequent syndrome.

We have set up a Data Safety Monitoring Board (DSMB) that will closely monitor the progress of the trial (DSMB Charter attached to this application). Any adverse event will be reported directly to the institutional review board (IRB) and DSMB. All adverse events will be reported in the annual review of the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Adults older than 18 years of age, admitted to the ICU with one or more of the following risk factors for ARDS/ALI:

  * Sepsis, defined as the presence of infection-related systemic inflammatory response syndrome (SIRS).

SIRS is defined as the presence of two or more of the following:

* Temperature >38.5ºC or <35ºC
* Heart rate >90 beats/min
* Respiratory rate >20 breaths/min or PaCO2 <32 mmHg
* WBC >12,000 cells/mm3, <4000 cells/mm3, or >10 percent immature (band) forms

  * Pneumonia, including community and health care associated pneumonias
  * Aspiration, defined as the witnessed inhalation of gastric contents
  * Acute pancreatitis
  * Bilateral lung contusion
  * Massive transfusion, defined as more than 15 units of red blood cells/24h
  * Multiple (>2) long-bone fractures

Exclusion Criteria:

* Patients already on a statin
* Current indication for statin therapy according to the National guidelines
* NPO order
* Active liver disease, defined as ALT or AST > 3 times the upper limits of normal
* History of myopathy
* History of uncontrolled seizure disorder
* Pregnancy or breastfeeding
* Immunosuppressive therapy, including prednisone at dose > 10 mg/day
* Preexistent lung disease indicated by history or chest film
* High risk for cardiogenic pulmonary edema (defined as the presence of ventricular fibrillation, acute myocardial infarction, congestive heart failure with EF < 40%)
* High risk for neurogenic pulmonary edema (active CVA, or known increased intracranial pressure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Incidence of ARDS/ALI. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jean Keddissi, M.D., Principal Investigator — University of Oklahoma; Gary T. Kinasewitz, MD, Principal Investigator — University of Oklahoma
Locations (2):
- United States (2):
  - OU Medical Center, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center, Oklahoma City, Oklahoma